CLINICAL TRIAL: NCT05560672
Title: Clinical Application and Mechanism of Cord Blood Mononuclear Cells in the Treatment of Ischemic Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YXLL-KY-2020(030)
Record Dates: First submitted 2022-09-20; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Bowel Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Cord blood mononuclear cell transplantation is performed at the same time as medical treatments such as fasting, rehydration, hemostasis, anti-infection, vasodilation, repair of intestinal mucosa, regulation of intestinal flora, etc.
  Interventions: Other: Human Umbilical Cord blood mononuclear cells
- Control group (No Intervention): Medical treatments such as fasting, rehydration, hemostasis, anti-infection, vasodilation, repair of intestinal mucosa, and regulation of intestinal flora are given.

INTERVENTIONS:
Other: Human Umbilical Cord blood mononuclear cells — Intravenous infusion of cord blood mononuclear cells
  Arms: Experimental group

SUMMARY:
Ischemic bowel disease, also known as ischemic bowel disease (IBD), is a type of disease that causes the blood supply to a certain intestinal segment to be reduced or stopped by various reasons such as hypovolemia, shock or recent abdominal surgery, resulting in insufficient blood supply to the intestinal wall, and causing a series of pathological changes in the intestine. Human umbilical cord blood mononuclear cells (HUCB-MNC) can be economically and conveniently isolated from human cord blood. The HUCB-MNC obtained from the isolation of human umbilical cord blood contains a variety of stem cells, such as hematopoietic stem cells, endothelial stem cells, etc. A number of previous studies have confirmed that HUCB-MNC can improve the occurrence of ischemic bowel disease through immunomodulatory and tissue repair. These characteristics make HUCB-MNC a cell with great potential to treat ischemic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age is not limited, gender is not limited. Meet the diagnostic criteria for ischemic bowel disease and clearly diagnose inpatient patients with ischemic bowel disease.
* Diagnosis and diagnosis (standard) in line with the "2011 Chinese Medical.
* Association Gerontology Branch organization of relevant experts jointly wrote the diagnosis and treatment of ischemic bowel disease in the elderly in China":

  1. Acute mesenteric ischemia (AMI): clinical manifestations are acute and severe abdominal pain, symptoms do not match the severity of signs, and signs are often not obvious. Abdominal x-ray may show "finger marks" and balloon signs. CT shows no visualization of the superior mesenteric artery or intraluminal filling defect. Arteriography is helpful in diagnosis, and intestinal mucosal pathology is dominated by ischemic changes, such as in patients with vasculitis, thrombosis, and vascular embolism.
  2. Chronic mesenteric ischemia (CMI): clinical symptoms are recurrent abdominal pain, chronic disease capacity, emaciation, no tenderness in the abdomen, and vascular murmurs can often be heard in the upper abdomen. Imaging tests such as arteriography, CTA, and MRA can help confirm the diagnosis of CMI. It is mainly based on clinical symptoms and advanced imaging tests.
  3. Ischemic colitis (IC): manifested as unexplained abdominal pain, bloody stool, diarrhea or abdominal acute abdomen, which can be diagnosed with colonoscopy and angiography if necessary.

Exclusion Criteria:

* The diagnosis does not conform to the "2011 Cases of Diagnosis and Treatment Recommendations for Ischemic Bowel Disease in the Elderly in China Jointly Written by Relevant Experts organized by the Geriatrics Branch of the Chinese Medical Association";
* Exclude those with serious diseases of other organs;
* Patients with other diseases such as gastrointestinal tumors and inflammatory bowel diseases cannot be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of IL-8 in serum | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after
  Ischemic bowel disease increases the expression of IL-8.
Concentration of NF-Kβ in serum | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after
  In the development of ischemic bowel disease, NFKβ activates the associated signaling pathway to exert an anti-inflammatory effect.
Concentration of IL-6 in serum | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after
  Ischemic bowel disease increases the expression of IL-6.
Concentration of IL-1β in serum | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after
  Ischemic bowel disease increases the expression of IL-1β.
Concentration of Nrf2 in serum | Compare the changes of 1 month, 3 months, 6 months and one year before treatment (baseline) and after
  In the development of ischemic bowel disease, Nrf2 interacts with NF-Kβ and has an anti-inflammatory effect.

CONTACTS AND LOCATIONS:
Locations (1):
- HongLi Yang, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No